CLINICAL TRIAL: NCT00636298
Title: Phase II Study of Cetuximab and Bevacizumab in Esophageal Carcinoma That Failed First Line Therapy
Brief Title: Study of Cetuximab and Bevacizumab in Cancer of the Esophagus After Failure of Patient's First Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Emory University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Nabil F. Saba, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006037; 6037 (Other: Other)
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Esophageal Carcinoma
Keywords: esophageal carcinoma; cancer of the esophagus; locally advanced or metastatic esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Single arm treatment with combination of cetuximab and bevacizumab
  Interventions: Drug: Bevacizumab, cetuximab

INTERVENTIONS:
Drug: Bevacizumab, cetuximab — Cetuximab - 400 mg/m2 loading, then 250 mg/m2 weekly
  Bevacizumab - 10 mg/kg every 2 weeks

SUMMARY:
The purpose of this study is to test the drug bevacizumab in combination with cetuximab. Because this combination has not been tested in cancer patients before, results will be analyzed to see what effects the combination of bevacizumab with cetuximab has on esophageal cancer.

DETAILED DESCRIPTION:
Cancer of the esophagus often has a poor outcome since many patients have advanced disease when they are diagnosed. The average survival rate after five years has increased from 4% in the 1970s to around 14% currently.

Surgery to remove the tumor or treatment with radiotherapy alone has led to disappointing results for patients. Chemotherapy has some activity in patients with advanced disease, although responses are usually short. New strategies are trying to combine these three treatment approaches to improve survival for these patients.

This study will test the combination of cetuximab and bevacizumab in patients with locally advanced esophageal cancer. This is a group of patients with usually poor outcomes from treatment with surgery, radiotherapy or chemotherapy alone. Scientifically, this study will help assess the value in combining these two different types of drug.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed squamous cell carcinoma or esophageal adenocarcinoma.
2. The disease must be recurrent after first line systemic therapy, with or without radiation, with or without surgery.
3. Patients must be at least 1 month from prior chemotherapy or radiation therapy.
4. ECOG performance status ≤ 1 (Karnofsky > 60%)
5. Life expectancy of greater than 12 weeks.
6. Age > 18.
7. Patients must have normal bone marrow and other organ function or defined below:

   * Absolute neutrophil count, > 1, 500/μL
   * Platelet counts, > 100, 00/μL

     _ Hemoglobin, > 8.0 gm/dL-
   * Creatinine(< 1.5mg/dL)
8. No significant intercurrent medical illness (including NYHA class II, III or IV heart disease, significant arrhythmias requiring medication, symptomatic coronary artery disease, myocardial infarction within the previous 6 months.
9. Women of childbearing potential must have a negative pregnancy test.
10. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

I. Disease-specific Exclusions

1. All histologic types other than squamous cell carcinoma or adenocarcinoma.
2. Patients currently receiving other investigational agents, or who have received cetuximab previously.
3. Patients with known brain metastases.
4. History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to Cetuximab or Bevacizumab.
5. Patients with history of any other malignancy (except non-melanomatous skin cancer or CIS of cervix) are ineligible unless a period of 5 years has lapsed since treatment of the previous cancer and the patient has remained continuously disease free.
6. Patients who are felt to be poorly compliant.
7. Women who are breast-feeding.

II. General Medical Exclusions

Subjects meeting any of the following criteria are ineligible for study entry:

1. Inability to comply with study and/or follow-up procedures.
2. Life expectancy of less than 12 weeks.
3. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study.

III. Bevacizumab-Specific Exclusions

1. Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure >100 mmHg on antihypertensive medications).
2. Any prior history of hypertensive crisis or hypertensive encephalopathy.
3. New York Heart Association (NYHA) Grade II or greater congestive heart failure
4. History of myocardial infarction or unstable angina within 6 months prior to study enrollment.
5. History of stroke or transient ischemic attack within 6 months prior to study enrollment.
6. Known CNS disease.
7. Significant vascular disease (e.g., aortic aneurysm, aortic dissection).
8. Symptomatic peripheral vascular disease.
9. Evidence of bleeding diathesis or coagulopathy.
10. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study.
11. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment.
12. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment.
13. Serious, non-healing wound, ulcer, or bone fracture.
14. Proteinuria at screening as demonstrated by either

    * Urine protein: creatinine (UPC) ratio ≥ 1.0 at screening OR
    * Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible)
15. Known hypersensitivity to any component of bevacizumab.
16. Pregnant (positive pregnancy test) or lactating. Use of effective means of contraception (men and women) in subjects of child-bearing potential.
17. History of myocardial infarction or unstable angina within 6 months of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Every 3 months

SECONDARY OUTCOMES:
Response rate | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Saba, MD, Principal Investigator — Emory University Winship Cancer Institute